CLINICAL TRIAL: NCT01071408
Title: Development of a Stroke Prevention Program for an Underserved Minority Community
Brief Title: Trial of a Secondary Stroke Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sepulveda Research Corporation (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Eric M. Cheng, Neurologist, Sepulveda Research Corporation
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: K23NS058571 (NIH); K23NS058571 (NIH)
Record Dates: First submitted 2010-02-12; First posted 2010-02-19 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: chronic care model; stroke prevention; health services research
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient | interventions — Chronic Care Model; Nurse Practitioners

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stroke Prevention Program + Usual Care (Experimental): Stroke Prevention Care Program + Usual Care. The Stroke prevention care program is in addition, not a substitute for usual care. Persons randomized to this arm are eligible to all care, including care by stroke specialists, while enrolled in the intervention.
  Interventions: Other: Stroke prevention care program
- Usual care (No Intervention)

INTERVENTIONS:
Other: Stroke prevention care program — Stroke prevention care program consists of group clinics, telephone coordination of care, and tracking of care through registries in the first 7 months after stroke or TIA presentation. A nurse practitioner will follow algorithms to adjust medications and to motivate patients to improve lifestyle habits.
  Other Names: group clinics; chronic care model; secondary stroke prevention program; nurse practitioner; medication algorithms
  Arms: Stroke Prevention Program + Usual Care

SUMMARY:
The purpose of this study is to determine whether an outpatient program can reduce the risk of recurrent stroke.

DETAILED DESCRIPTION:
Stroke is a major cause of death and disability. A history of stroke is the strongest predictor of a future stroke. Control of risk factors lowers the risk of future stroke, yet most persons with stroke do not have their risk factors controlled.

In this randomized-controlled trial, we will test whether an outpatient stroke prevention program consisting of group clinics, patient self-management, and telephone care coordination can lower the risk of recurrent stroke by improving patient knowledge, medication adherence, and lifestyle habits. If successful, this program may be adapted to other settings.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke within the past 30 days
* transient ischemic attack within the past 30 days
* person receiving care at VA Long Beach Healthcare System

Exclusion Criteria:

* unable to understand informed consent
* already enrolled in another research study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Blood pressure control | baseline, 3 months, 7 months

SECONDARY OUTCOMES:
control of other stroke risk factors including lipids, smoking, and exercise | baseline, 3 months, 7 months
patient perceptions of care quality | baseline, 3 months, 7 months
medication adherence | baseline, 3 months, 7 months
Stroke knowledge | baseline, 3 months, 7 months
  Open ended questions about the warning signs about stroke. Open ended questions about the risk factors of stroke. These questions evaluate the effectiveness of the didactic portion of the group sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Cheng, MD, MS, Principal Investigator — VA Long Beach Healthcare System
Locations (1):
- VA Long Beach Health Care System, Long Beach, California, United States